CLINICAL TRIAL: NCT00751231
Title: A Randomized, Double-Blind, Active-Controlled Trial to Evaluate Intravenous and Oral PRT060128, a Selective and Reversible P2Y12 Inhibitor, vs Clopidogrel, as a Novel Antiplatelet Therapy in Patients Undergoing Non-Urgent PCI
Brief Title: A Phase 2 Safety and Efficacy Study of PRT060128, a Novel Intravenous and Oral P2Y12 Inhibitor, in Non-Urgent PCI
Acronym: INNOVATE-PCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-116; 2008-001352-51 (EudraCT Number)
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Percutaneous Coronary Intervention
Keywords: PCI; percutaneous coronary intervention
MeSH Terms: interventions — Clopidogrel; elinogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Active Comparator): 300mg or 600mg loading dose of Clopidogrel followed by once daily dosing of 75 mg Clopidogrel for up to 120 days.
  Interventions: Drug: clopidogrel
- Arm 2 (Experimental): IV bolus of PRT060128 prior to PCI and twice daily administration of 50 mg oral PRT060128 for up to 120 days, with the first oral dose administered concurrently with the IV bolus.
  Interventions: Drug: PRT060128
- Arm 3 (Experimental): IV bolus of PRT060128 prior to PCI and twice daily administration of 100 mg oral PRT060128 for up to 120 days, with the first oral dose administered concurrently with the IV bolus.
  Interventions: Drug: PRT060128
- Arm 4 (Experimental): IV bolus of PRT060128 prior to PCI and twice daily administration of 150 mg oral PRT060128 for up to 120 days, with the first oral dose administered concurrently with the IV bolus.
  Interventions: Drug: PRT060128

INTERVENTIONS:
Drug: clopidogrel — Loading dose of 300mg or 600mg, followed by once daily dosing of 75 mg
  Other Names: Plavix
  Arms: Arm 1
Drug: PRT060128 — 80-120 mg IV bolus administered prior to PCI, followed by twice daily dosing of oral 50mg, 100mg or 150mg
  Arms: Arm 2; Arm 3; Arm 4

SUMMARY:
This is a multi-center, randomized, double-blind, triple-dummy, clopidogrel-controlled study of IV and oral PRT060128 compared to clopidogrel in patients undergoing non-urgent (including elective) PCI. After diagnostic angiography, patients scheduled for non-urgent PCI will be randomized to clopidogrel or to one of three dose levels of PRT060128.

DETAILED DESCRIPTION:
Each patient randomized in this trial will participate for approximately 12-24 weeks, including a Screening period of up to 2 weeks, the acute peri-procedural phase, and a 60-120 day chronic treatment phase. The chronic phase includes daily in-hospital assessments until 24 Hours or Discharge (whichever comes first), a telephone follow-up on Day 7-10 post-Discharge, outpatient follow-up visits on Days 30 and 60-67, [Day 90 and Day 120 (if treated for 120 days)] and a telephone follow-up 7 days following the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* The patient is scheduled to undergo non-urgent PCI
* The patient is between 18 and 75 years of age (inclusive) and willing to comply with the protocol
* Women of childbearing potential must have a negative serum or urine pregnancy test within 24 hours of dosing. All patients must agree to use double barrier contraception during the study and for at least 4 weeks after their last dose.
* The patient or legally acceptable representative is able to read and give written informed consent and has signed an informed consent form approved by the Investigator's IRB/IEC

Exclusion Criteria:

* Estimated or measured weight < 55 kg
* Acute non-ST-segment elevation myocardial infarction (NSTEMI) or ST-segment elevation myocardial infarction (STEMI) within 7 days prior to PCI
* Chronic total occlusion or unprotected left main stenting
* Cardiogenic shock (systolic blood pressure < 90 mm Hg requiring vasopressor or hemodynamic support)
* Uncontrolled hypertension at the time of initial study drug administration defined as measured systolic blood pressure > 190 mm Hg or diastolic blood pressure > 108 mm Hg
* Planned staged PCI
* Planned surgery during the study period
* Planned GP IIb/IIIa use
* Patient has received a clopidogrel loading dose (≥300 mg) within 7 days prior to randomization; patients on maintenance clopidogrel may be enrolled
* The planned administration of the study-specified clopidogrel loading dose is >12 hours prior to PCI
* Administration of thrombolytic agents, fondaparinux, or oral anticoagulants (e.g., warfarin) within the 7 days prior to PCI
* Estimated creatinine clearance (e.g. Cockcroft-Gault) < 45 mL/min
* Anemia with hemoglobin level < 10 g/dL
* Thrombocytopenia (platelet count < 100,000/mm3)
* ALT and/or AST > 2.5 x the ULN or other indication of clinically significant hepatic dysfunction
* Facial or head trauma within the last 30 days
* Intraocular hemorrhage within the last 30 days
* Gastrointestinal bleeding within the last 30 days
* Active bleeding, or history of a bleeding disorder or known intracranial vascular malformation
* History of any prior ischemic stroke or TIA within the last 5 years or intracranial hemorrhage, neoplasm, or arteriovenous malformation
* Known allergy or contraindication to the components of PRT060128, aspirin, heparin, clopidogrel, glycoprotein IIb/IIIa inhibitors, or to any contrast media
* Participation in any investigational drug study within 30 days prior to enrollment. Participation in a device trial prior to enrollment is acceptable
* Prior participation in any study involving PRT060128
* Any condition which could interfere with, or the treatment for which might interfere with, the conduct of the study or which would, in the opinion of the Investigator, unacceptably increase the patient's risk by participating in the study. This would include, but is not limited to alcoholism, drug dependency or abuse, psychiatric disease, epilepsy or any unexplained blackouts

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The study is not powered to examine a pre-specified endpoint; rather it is designed to explore a number of analyses to understand the clinical efficacy, biological activity, and tolerability and safety of PRT060128 in patients undergoing non-urgent PCI | 24 Hours/Discharge and Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Robert Harrington, MD, Study Chair — Duke University; Sunil V Rao, MD, Principal Investigator — Duke University; Robert C Welsh, MD, Principal Investigator — University of Alberta
Locations (59):
- United States (19):
  - Portola Investigational Site, La Jolla, California
  - Portola Investigational Site, Torrance, California
  - Portola Investigational Site, Washington D.C., District of Columbia
  - Portola Investigational Site, Jacksonville, Florida
  - Portola Investigational Site, Tallahassee, Florida
  - Portola Investigational Site, Augusta, Georgia
  - Portola Investigational Site, Lexington, Kentucky
  - Portola Investigational Site, New Orleans, Louisiana
  - Portola Investigational Site, Portland, Maine
  - Portola Investigational Site, Baltimore, Maryland
  - Portola Investigational Site, Detroit, Michigan
  - Portola Investigational Site, Grand Blanc, Michigan
  - Portola Investigational Site, Brooklyn, New York
  - Portola Investigational Site, Charleston, North Carolina
  - Portola Investigational Site, Winston-Salem, North Carolina
  - Portola Investigational Site, Cincinnati, Ohio
  - Portola Investigational Site, Hershey, Pennsylvania
  - Portola Investigational Site, Lancaster, Pennsylvania
  - Portola Investigational Site, Seattle, Washington
- Austria (2):
  - Portola Investigational Site, Graz
  - Portola Investigational Site, Vienna
- Canada (6):
  - Portola Investigational Site, Calgary, Alberta
  - Portola Investigational Site, Edmonton, Alberta
  - Portola Investigational Site, Vancouver, British Columbia
  - Portola Investigational Site, St. John's, Newfoundland and Labrador
  - Portola Investigational Site, Newmarket, Ontario
  - Portola Investigational Site, Toronto, Ontario
- Germany (26):
  - Portola Investigational Site, Bad Oeynhausen
  - Portola Investigational Site, Bad Rothenfelde
  - Portola Investigational Site, Berlin
  - Portola Investigational Site, Bernau
  - Portola Investigational Site, Dachau
  - Portola Investigational Site, Dortmund
  - Portola Investigational Site, Dresden
  - Portola Investigational Site, Göttingen
  - Portola Investigational Site, Halle
  - Portola Investigational Site, Hanover
  - Portola Investigational Site, Heidelberg
  - Portola Investigational Site, Kassel
  - Portola Investigational Site, Kiel
  - Portola Investigational Site, Langen
  - Portola Investigational Site, Ludwigshafen
  - Portola Investigational Site, Lübeck
  - Portola Investigational Site, Mainz
  - Portola Investigational Site, Mönchengladbach
  - Portola Investigational Site, Munich
  - Portola Investigational Site, Neuss
  - Portola Investigational Site, Rostock
  - Portola Investigational Site, Schwalmstadt
  - Portola Investigational Site, Traunstein
  - Portola Investigational Site, Trier
  - Portola Investigational Site, Witten
  - Portola Investigational Site, Wuppertal
- Poland (6):
  - Portola Investigational Site, Bydgoszcz
  - Portola Investigational Site, Gdansk
  - Portola Investigational Site, Lodz
  - Portola Investigational Site, Lublin
  - Portola Investigational Site, Szczecin
  - Portola Investigational Site, Warsaw

REFERENCES:
- [Derived] Welsh RC, Rao SV, Zeymer U, Thompson VP, Huber K, Kochman J, McClure MW, Gretler DD, Bhatt DL, Gibson CM, Angiolillo DJ, Gurbel PA, Berdan LG, Paynter G, Leonardi S, Madan M, French WJ, Harrington RA; INNOVATE-PCI Investigators. A randomized, double-blind, active-controlled phase 2 trial to evaluate a novel selective and reversible intravenous and oral P2Y12 inhibitor elinogrel versus clopidogrel in patients undergoing nonurgent percutaneous coronary intervention: the INNOVATE-PCI trial. Circ Cardiovasc Interv. 2012 Jun;5(3):336-46. doi: 10.1161/CIRCINTERVENTIONS.111.964197. Epub 2012 May 29. PMID 22647518
- [Derived] Angiolillo DJ, Welsh RC, Trenk D, Neumann FJ, Conley PB, McClure MW, Stephens G, Kochman J, Jennings LK, Gurbel PA, Wojcik J, Dabrowski M, Saucedo JF, Stumpf J, Buerke M, Broderick S, Harrington RA, Rao SV. Pharmacokinetic and pharmacodynamic effects of elinogrel: results of the platelet function substudy from the intravenous and oral administration of elinogrel to evaluate tolerability and efficacy in nonurgent percutaneous coronary intervention patients (INNOVATE-PCI) trial. Circ Cardiovasc Interv. 2012 Jun;5(3):347-56. doi: 10.1161/CIRCINTERVENTIONS.111.965608. Epub 2012 May 22. PMID 22619259
- See also: A Randomized, Double-Blind, Active-Controlled Phase 2 Trial to Evaluate a Novel Selective and Reversible Intravenous and Oral P2Y12 Inhibitor Elinogrel Versus Clopidogrel in Patients Undergoing Nonurgent PCI: The INNOVATE-PCI Trial — http://www.ncbi.nlm.nih.gov/pubmed/22647518
- See also: Pharmacokinetic and Pharmacodynamic Effects of Elinogrel: Results of the Platelet Function Substudy From the Intravenous and Oral Administration of Elinogrel to Evaluate Tolerability and Efficacy in Nonurgent PCI Patients (INNOVATE-PCI) Trial — http://www.ncbi.nlm.nih.gov/pubmed/22619259